CLINICAL TRIAL: NCT06200597
Title: A Phase 1 Randomized, 2-part, Single-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of LAD603 in Healthy Adult Subjects
Brief Title: A Single and Multiple Ascending Dose Study of LAD603 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-00223-01
Record Dates: First submitted 2023-12-22; First posted 2024-01-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part 1: (LAD603) Cohort 1 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 2 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 3 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 4 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 5 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 6 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 7 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: (LAD603) Cohort 8 (Experimental): Participants will receive single ascending dose of LAD603 SC injection on Day 1.
  Interventions: Drug: LAD603
- Part 1: Placebo (Placebo Comparator): Participants will receive single ascending dose of matching placebo SC injection on Day 1.
  Interventions: Other: Placebo
- Part 2: (LAD603) Cohort A (Experimental): Participants will receive multiple ascending dose of LAD603 SC injection on Days 1, 15, 18 and 22.
  Interventions: Drug: LAD603
- Part 2: (LAD603) Cohort B (Experimental): Participants will receive multiple ascending dose of LAD603 SC injection on Days 1, 15, 18 and 22.
  Interventions: Drug: LAD603
- Part 2: (LAD603) Cohort C (Experimental): Participants will receive multiple ascending dose of LAD603 SC injection on Days 1, 15, 18 and 22.
  Interventions: Drug: LAD603
- Part 2: (LAD603) Cohort D (Experimental): Participants will receive multiple ascending dose of LAD603 SC injection on Days 1, 15, 18 and 22.
  Interventions: Drug: LAD603
- Part 2: Placebo (Placebo Comparator): Participants will receive multiple ascending dose of matching placebo SC injection on Days 1, 8 15, and 22.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LAD603 — LAD603 SC injection.
  Arms: Part 1: (LAD603) Cohort 1; Part 1: (LAD603) Cohort 2; Part 1: (LAD603) Cohort 3; Part 1: (LAD603) Cohort 4; Part 1: (LAD603) Cohort 5; Part 1: (LAD603) Cohort 6; Part 1: (LAD603) Cohort 7; Part 1: (LAD603) Cohort 8; Part 2: (LAD603) Cohort A; Part 2: (LAD603) Cohort B; Part 2: (LAD603) Cohort C; Part 2: (LAD603) Cohort D
Other: Placebo — Matching placebo SC injection.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single and multiple ascending doses of LAD603 in healthy adult participants in both Part 1 and 2.

DETAILED DESCRIPTION:
This is a 2-part study. Part 1 will comprise up to 8 cohorts of healthy adult participants and investigate single ascending doses of LAD603. Part 2 will comprise up to 4 cohorts of healthy adult subjects and will investigate multiple ascending doses of LAD603. Each ascending dose level will be investigated by a sequential cohort, with dose escalation based on satisfactory safety, tolerability, PK, and pharmacodynamics (PD) (biomarker) data from the previous cohort(s). Dose levels evaluated in Part 2 of this study will not exceed dose levels that were safe and well tolerated in the single-dose study, and may be changed, depending on emerging safety and tolerability, PK, and PD (biomarker) data.

Each participant will participate for about 8 weeks in Part 1 and for about 14 weeks in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male or female aged between 18 and 65 years, inclusive, at the time of signing the informed consent.
2. Participant is willing and able to understand and comply with study requirements
3. Participant is willing to participate and have provided signed informed consent in accordance with institutional and regulatory guidelines, and authorization to use protected health information (Health Insurance Portability and Accountability Act [HIPAA]) prior to any study-related procedures being performed.
4. Participant has a body mass index (BMI) of greater than or equal to (>=) 18.5 and less than or equal to (<=) 29.9 kilogram per meter square (kg/m^2) with a body weight of at least 60 kg.
5. Participant is in good health as determined by medical history and has no clinically relevant abnormalities in the physical examination, vital signs, 12-lead ECG, and laboratory tests as determined by the Investigator.
6. Participant is a female who is not pregnant (i.e., does not have a positive serum pregnancy test on Day -1]) or breastfeeding, and who is either not a WOCBP or is a WOCBP who agrees to follow the contraceptive guidance for at least 28 days or 1 menstrual period (whichever is longer) prior to Day -1 until 30 days after the last dose of investigational medical product (IMP) and to refrain from egg donation/collection until at least 60 days after the last dose of IMP OR Participant is a male who either had a vasectomy at least 90 days prior to Screening (with appropriate post vasectomy documentation of absence of sperm in the ejaculate) or who agrees to use contraception from the Day 1 visit until 30 days after the last dose of IMP and to refrain from sperm donation during this period, or is a vasectomized male who agrees to use a condom from the Day 1 visit until 30 days after the last dose of IMP.

Exclusion Criteria:

1. Participant has a history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, inflammatory, or allergic disease (including drug allergies, any active seizure disorder requiring therapy with antiepileptic drugs, active peptic ulcer disease, gastrointestinal bleeding, chronic gastritis, inflammatory bowel disease or chronic diarrhea, but excluding mild seasonal allergies or stable, well-controlled thyroiditis), a history of organ transplant, or is at increased risk for capillary leak syndrome.
2. Participant has had major surgery (requiring general anesthesia) within 3 months prior to Baseline (Day -1).
3. Participant has a history of cancer or lymphoproliferative disease within the previous 5 years, other than resected cutaneous basal cell, squamous cell carcinoma or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
4. Participant has a clinically significant ECG abnormality at Screening or Baseline (Day -1), including, but not limited to, the following:

   * An abnormal PR interval (>=220 millisecond [msec] or <=100 msec)
   * QTc prolongation (corrected QT interval by Fredericia's formula [QTcF] >=450 msec)
5. Participant has a mean heart rate (HR) at Screening or Baseline (Day -1) that is <=45 beats per minute (bpm) or >100 bpm
6. Participant has systolic blood pressure <90 millimeter of mercury (mmHg) or >140 mmHg or diastolic blood pressure <50 mmHg or >90 mmHg at Screening or Baseline (Day -1)
7. Participant with active chronic or acute infection including skin infection requiring treatment with systemic antimicrobials, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before Baseline (Day -1), or skin infections within 4 weeks prior to Baseline (Day -1), or fever >38°C of unknown etiology within 1 week prior to Baseline (Day -1).
8. Participant has known hypersensitivity to any of the formulation excipients of the IMP or previous severe adverse reaction to subcutaneous medication.
9. Participant has hypersensitivity or reaction to a prior antibody-based biologic therapy (regardless of indication) that was clinically significant, as per judgment of Investigator.
10. Participant has positive results for hepatitis B surface antigen (HBsAg), antihepatitis B core antigen (anti-HBcAg), antibody to the hepatitis C virus (anti-HCV), or antibody to the human immunodeficiency virus (HIV-1/2). A history of hepatitis B vaccination without history of hepatitis B is allowed.
11. Participant has a positive test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) prior to dosing at Baseline (Day -1).
12. Participant has received any type of live or attenuated vaccinations within 28 days prior to Baseline (Day -1), or is planning to receive any such vaccine during the study (inactive vaccines are allowed) or has received a SARS-CoV-2 vaccine within 14 days prior to Baseline (Day -1). Seasonal influenza and H1N1 vaccinations are permitted if the inactivated vaccine formulation is administered.
13. Participant with history of active or latent tuberculosis, or recent close contact with an individual with active tuberculosis, or is positive at the Screening visit by tuberculin blood test (eg, QuantiFERON).
14. Participant with congenital or acquired immunosuppressive condition that would put participant at risk during the study.
15. Participant with a history (within 6 months prior to Screening visit) of drug and/or alcohol abuse that may prevent trial compliance based on Investigator judgment.
16. Females who are pregnant or breast-feeding or seeking to become pregnant during the study or for approximately 30 days after the last dose of IMP.
17. Participant is a current smoker and is unable to restrain from smoking during the study.
18. Participant has a positive test for drugs of abuse and/or alcohol.
19. Participant has received any investigational drug in any clinical study within 30 days (or at least 5 half-lives, whichever is longer) prior to Baseline (Day -1) or is on extended follow-up from such a clinical study
20. Participant has taken any medications, including over-the-counter (OTC) medications, within 14 days (or at least 5 half-lives, whichever is longer) before Baseline (Day -1) (note that hormonal contraceptives are allowed, and acetaminophen is permitted at doses <=2 gram per day (g/day) up to 48 hours prior to each study visit), unless in the opinion of the Investigator and CRO Medical Monitor the medication will not interfere with the study procedures or compromise participant safety. Participants taking drugs that are substrates of cytochrome P450 or have a narrow therapeutic index are excluded from participating in this study.
21. Participants with ANY of the following abnormalities in clinical laboratory tests at Screening or, if applicable, Day -1, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

    * Neutrophil or lymphocyte counts below the lower limit of the normal range.
    * Eosinophil count above the normal range (i.e., >500/mm^3).
    * Estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation <=90 mL/min/1.73 m^2 at Screening.
    * Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) or alkaline phosphatase (ALP) > Upper limit of the normal range (ULN).
    * Total bilirubin >ULN
    * Other clinically significant abnormalities of laboratory assessments, as judged by the Investigator and/or Sponsor Medical Monitor that could affect the safety of the participant, or the interpretation of the data from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) and Severity of AEs | Baseline up to Day 31
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Vital Sign Parameter | Baseline up to Day 31
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Electrocardiograms (ECGs) Parameters | Baseline up to Day 31
Part 1: Number of Participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | Baseline up to Day 31
Part 2: Number of Participants with AEs and Severity of AEs | Baseline up to Day 64
Part 2: Number of Participants with Clinically Significant Changes from Baseline in Vital Sign Parameter | Baseline up to Day 64
Part 2: Number of Participants with Clinically Significant Changes from Baseline in ECGs Parameters | Baseline up to Day 64
Part 2: Number of Participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | Baseline up to Day 64

SECONDARY OUTCOMES:
Part 1: Maximum Serum Concentration (Cmax) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Minimum Serum Concentration (Cmin) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Time to Reach Maximum Serum Concentration (Tmax) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Area Under the Serum Concentration-time Curve (AUC) from Zero to Time of the Last Concentration (AUC0-t) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Area Under the Serum Concentration-time Curve (AUC) from Zero to infinity (AUC0-inf) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Area Under the Serum Concentration-time Curve (AUC) from Zero to 1 Week After Investigational Medicinal Product (IMP) Administration (AUC0-1w) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Elimination Half-life (t½) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Smallest Terminal Elimination Rate Constant (λz) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Apparent Total Serum Clearance (CL/F) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Mean Residence Time (MRT) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 1: Apparent Volume of Distribution Associated with the Terminal Phase (Vz/F) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: at 24 and 36 hours (Day 2), 48 hours (Day 3), 72 hours (Day 4), 120 hours (Day 6), 168 hours (Day 8), 240 hours (Day 11); 336 hours (Day 15), 504 hours (Day 22), 672 hours (Day 29)
Part 2: Area Under the Concentration-time Curve within a Dosing Interval (AUCτ) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 1)
Part 2: Maximum Serum Concentration (Cmax) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 1)
Part 2: Time to Reach Maximum Serum Concentration (Tmax) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Area Under the Concentration-time Curve within a Dosing Interval (AUCτ) at Steady State of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Average Steady State Serum Drug Concentration (Cav,ss) | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Elimination Half-life (t½) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Smallest Terminal Elimination Rate Constant (λz) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Accumulation Ratios (RA) at Steady State Based on AUCτ (RA[AUC]) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Accumulation Ratios (RA) at Steady State Based on Cmax (RA[Cmax]) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Serum Concentration Observed at the Last Planned Sampling Timepoint Prior to Dosing (Ctrough; RA[Ctrough]) of LAD603 | Pre-dose, 2, 6, and 12 hours post-dose (Day 22)
Part 2: Serum Concentration Observed at the Last Planned Sampling Timepoint Prior to Dosing (Ctrough) of LAD603 | Pre-dose, 2, 6, 12 hours (Day 1); Post-dose: 24 and 36 hours (Day 2), 48 hours (Day 3), 96 hours (Day 5), 168 hours (Day 8); Pre-dose (Day 15); Pre-dose, 2, 6, and 12 hours post-dose (Day 22)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Phase 1 unit Lenexa, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR